CLINICAL TRIAL: NCT01569100
Title: Atorvastatin Effect in Incidence and Ischemic Complications of Vasospasm After Subarachnoid Aneurysmal Hemorrhage: a Cohort Study
Brief Title: Atorvastatin After Aneurysmal Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Louis Puybasset, Professor, Chief of the Intensive Care Neurosurgical Unit, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: REASTAT01
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: SAH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors, known as statins, have recently been demonstrated to improve endothelial function. Additionally, numerous studies have shown statins as having antiinflammatory and cell-signaling effects together with a selective up-regulation of the eNOS activity. These findings are of potential benefit for the prevention of cerebral vasospasm after a aneurysmal subarachnoid hemorrhage. Indeed, one of the possible mechanisms for this vasospasm is the eNOS depletion or even increase of eNOS expression after the hemorrhage. The purpose of this study is to observe the immediate effect of statins after aneurysmal subarachnoid hemorrhage (aSAH) in cerebral vasospasm and outcome at one year.

DETAILED DESCRIPTION:
Up to now, the preventive and curative treatment of vasospasm secondary to subarachnoid aneurismal hemorrhage has been based on three major approaches: increasing arterial pressure and cerebral blood flow with the use of triple H therapy, increasing the ischemic threshold of neurons with nimodipine and reopening proximal arteries with angioplasty and/or intra-arterial administration of nimodipine, verapamil, milrinone or papaverine. Recently, several teams have observed the efficacy of diverse statins in the prevention of vasospasm by improving the imbalance between the nitric oxide and the endothelin pathways, a major actor in the physiopathology of vasospasm. Indeed, this family of molecules improve the bioavailability of endogenous nitric oxide and upregulate the endothelial NO synthase.

In humans, statin administered within the first 72 hours showed to significantly reduce the incidence of vasospasm up to 50% an therefore, induce a lower morbidity and mortality of this severely ill population. The aim of this study is to demonstrate that atorvastatin reduces the incidence of cerebral vasospasm-related morbidity and mortality within 1 year post aneurysmal subarachnoid hemorrhage (aSAH) treated by either clipping or endovascular coiling.

ELIGIBILITY:
Inclusion Criteria:

* SAH patient > 16 years-old admitted to the Pitie- Salpetriere Teaching Hospital
* Securing procedure within 96 hours of bleeding

Exclusion Criteria:

* Securing procedure > 96 hours of bleeding
* Rebleeding of original aneurysm

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted between April 20, 2004, and October 1, 2007, to the Pitie- Salpetriere Teaching Hospital in Paris with aneurysmal SAH and treated by endovascular coiling or surgery within 96 hrs after SAH onset were considered for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
S100B assay measured daily from days 1-15 | Day 1 through 15

SECONDARY OUTCOMES:
Ischemic lesion volume | admission upon death or hospital discharge
  Ischemic lesion voulume was measured on the last available CT prior to death or hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Louis Puybasset, Pr, Principal Investigator — Departments of Anesthesiology and Critical Care, Pitie-Salpetriere Hospital, APHP, University Pierre et Marie Curie, Paris, France